CLINICAL TRIAL: NCT02221453
Title: Cytokine Levels in Patients With Persistent Diabetic Macular Edema Treated With Triamcinolone Acetonide: an Interventional Prospective Study
Brief Title: Cytokine Levels in Patients With Persistent Diabetic Macular Edema Treated With Triamcinolone Acetonide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PersDMEcytokineTA
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Ocular Cytokines; Triamcinolone Acetonide
MeSH Terms: interventions — Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triamcinolone Acetonide Treatment (Other): Triamcinolone Acetonide Injectable Suspension 40 mg/mL intravitreal injection
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide
  Other Names: Triesence

SUMMARY:
Diabetic macular edema refers to swelling (fluid accumulation) in the center of the retina. The retina is like the film of a camera and is located in the back of the eye. This condition can develop in diabetics where swelling results from leaking of fluid from the blood vessels of the eye, into the center of the retina, the macula. If left untreated, this can affect central vision. The current standard treatment for diabetic macular edema includes medications injected directly into the eye (intravitreal injections) and laser eye treatment. The drugs that are injected directly into the eye are known as anti-Vascular Endothelial Growth Factor (anti-VEGF) agents which help to reduce the leaking. This includes bevacizumab (Avastin®) and ranibizumab (Lucentis®).

However, some patients do not respond well to these anti-VEGF treatments will be given the option of switching to an another class of medications, called steroids. Triamcinolone acetonide is one of these steroids and is also injected directly into the eye. These steroids will help reduce inflammation and possibly as a consequence, reduce swelling in the eye.

The purpose of this study is to determine what cellular factors affect a patient's treatment response (amount of swelling reduction) following triamcinolone acetonide intravitreal injections for diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Non Proliferative Diabetic Retinopathy (NDPR) or Proliferative Diabetic Retinopathy as confirmed by IntraVenous Fluorescein Angiography (IVFA)
* Prior treatment with ≥ 6 intravitreal anti-VEGF injections but no treatment in last 4 weeks
* Less than 10% improvement in Central Macular Thickness on OCT scan and less than 1 line improvement in vision from baseline
* Less than 10% reduction in macular volume
* Age 18 years or older
* Subjects with Type I or II diabetes mellitus
* snellen Acuity 20/40 to 20/400 and its ETDRS equivalent
* Ability to provide signed informed consent
* Capable of complying with study protocol.

Exclusion Criteria:

* Previous intraocular injection of steroid medication.
* Concurrent ocular disease (wet Age-Related Macular Degeneration, significant Epiretinal Membrane, vitreomacular traction etc) that would limit visual acuity in the opinion of the treating physician
* Proliferative diabetic retinopathy in the study eye or PanRetinal Photocoagulation within the last 12 months
* Poor glycemic control HbA1c >9%
* Prior vitrectomy surgery.
* Prior intraocular surgery within 3 months in study eye
* Laser treatment within 3 months of study eye
* Use of systemic steroids (eg, oral, intravenous, intramuscular, epidural, rectal, or extensive dermal) within 1 month prior to study enrollment.
* Known history of Intraocular Pressure (IOP) elevation in response to steroid treatment in either eye that resulted in any of the following: a) = 10 mm Hg increase in IOP in response to steroid injection, or b) IOP = 25 mm Hg and required 2 or more anti-glaucoma medications to keep IOP below 21 mm Hg.
* Known allergies to study drug or fluorescein
* History of stroke or acute Myocardial Infarction within 6 months of enrolment
* Patients receiving dialysis for renal failure
* Patients currently on systemic immunosuppression
* Patients with glaucoma
* Patients who are pregnant.
* Unwilling or unable to follow or comply with all study related procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in cytokine levels (picograms per mL) between baseline triamcinolone acetonide injection and 3 months | 3 months after baseline triamcinolone acetonide injection
  The study involves the measurement of ocular cytokines in the anterior chamber fluid including: EGF, VEGF, PlGF, IL-2, IL-3, IL-6, IL-17, TGF-B2, IL-8, VCAM, TGF-B, MMP-9, MIG, ICAM-1 and MCP-1.
Change in cytokine levels (picograms per mL) 3 months after 2nd triamcinolone acetonide injection | 3 months after 2nd triamcinolone acetonide injection
  Note that the 2nd triamcinolone acetonide injection occurs 3 months after baseline injection. The study involves the measurement of ocular cytokines in the anterior chamber fluid including: EGF, VEGF, PlGF, IL-2, IL-3, IL-6, IL-17, TGF-B2, IL-8, VCAM, TGF-B, MMP-9, MIG, ICAM-1 and MCP-1.

SECONDARY OUTCOMES:
Change in ocular cytokine levels (picograms per mL) in relation to change in Early Treatment of Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) in response to steroid treatment | 3 months after baseline injection
  The study involves the measurement of ocular cytokines in the anterior chamber fluid including: EGF, VEGF, PlGF, IL-2, IL-3, IL-6, IL-17, TGF-B2, IL-8, VCAM, TGF-B, MMP-9, MIG, ICAM-1 and MCP-1. Change in ETDRS BCVA is in ETDRS letters.
Change in ocular cytokine levels (picograms per mL) in relation to change in Early Treatment of Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) in response to steroid treatment | 3 months after 2nd triamcinolone acetonide injection
  The study involves the measurement of ocular cytokines in the anterior chamber fluid including: EGF, VEGF, PlGF, IL-2, IL-3, IL-6, IL-17, TGF-B2, IL-8, VCAM, TGF-B, MMP-9, MIG, ICAM-1 and MCP-1. Change in ETDRS BCVA is in ETDRS letters.
Change in ocular cytokine levels (picograms per mL) in relation to change in central macular thickness (CMT) measured in micrometers (um) from optical coherence tomography | 3 months after baseline injection
  The study involves the measurement of ocular cytokines in the anterior chamber fluid including: EGF, VEGF, PlGF, IL-2, IL-3, IL-6, IL-17, TGF-B2, IL-8, VCAM, TGF-B, MMP-9, MIG, ICAM-1 and MCP-1. Change in CMT is in micrometers (um).
Change in ocular cytokine levels (picograms per mL) in relation to change in central macular thickness (CMT) measured in micrometers (um) from optical coherence tomography | 3 months after 2nd triamcinolone acetonide injection
  The study involves the measurement of ocular cytokines in the anterior chamber fluid including: EGF, VEGF, PlGF, IL-2, IL-3, IL-6, IL-17, TGF-B2, IL-8, VCAM, TGF-B, MMP-9, MIG, ICAM-1 and MCP-1. Change in CMT is in micrometers (um).

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Muni, MD MSc FRCSC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital Eye Clinic, Toronto, Ontario, Canada